CLINICAL TRIAL: NCT04983498
Title: Evaluation of an Enhanced Recovery Pathway for Endoscopy Patients Receiving Moderate Sedation
Brief Title: Enhanced Recovery Pathway for Endoscopy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator left organization before study initiated.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Angela Maeder, PhD, RNC-OB, Clinical Nurse, Labor and Delivery Northwestern Memorial Hospital, Northwestern University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: STU00214245
Record Dates: First submitted 2021-07-20; First posted 2021-07-30 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Enhanced Recovery Pathway; Endoscopy
MeSH Terms: interventions — Ondansetron; Ringer's Lactate; Early Ambulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prospective Experimental Group (Experimental): For the experimental group, we will recruit 200 participants who will receive the Enhanced Recovery Pathway, which will be ordered as a standing order set by the attending provider and managed by their peri-procedural nurses. The modified ERP for this study includes the following interventions: nursing managed order sets with ERP instructions to receive goal-directed fluid management within anesthesia approved parameters utilizing the NMH Colorectal ERAS protocol for IV fluid administration, PONV prophylaxis for participants with an apfel score of 2 or greater (ondansetron 4 mg IV), an additional dose of ondansetron 4mg IV will be available in recovery if the patient has nausea/vomiting despite prophylaxis, early mobilization up to chair (within 5-30 minutes of admission to the recovery room) based on nursing parameters, and early PO intake within 15-30 minutes of admission to the recovery room post-procedure based on nursing parameters.
  Interventions: Drug: Ondansetron 4 MG; Drug: Lactated Ringers, Intravenous; Other: Early Mobilization; Other: Early PO Intake
- Retrospective Control Group (No Intervention): The retrospective group will consist of 200 randomly selected medical records of patients who had colonoscopy procedures for a 6 month period prior to study implementation (between 10/1/2019 to 4/1/2020). The retrospective control group will have received the current standard of care including: IV fluids for management of intra-procedural hypotension as indicated/ordered by the physician, PO intake at 30-45 minutes, up to a chair at 60 minutes, and all procedure related complications will have been treated (e.g. PONV) per physician order as is the current standard of practice in the GI Lab recovery area.

INTERVENTIONS:
Drug: Ondansetron 4 MG — PONV prophylaxis for participants with an apfel score of 2 or greater (ondansetron 4 mg IV), an additional dose of ondansetron 4mg IV will be available in recovery if the patient has nausea/vomiting despite prophylaxis.
  Other Names: Post-operative Nausea & Vomiting Prophylaxis
  Arms: Prospective Experimental Group
Drug: Lactated Ringers, Intravenous — Goal directed IV fluids to be administered starting preop per the NMH Colorectal ERAS protocol (LR @ 5mL/kg/hr).
  Other Names: Intravenous Hydration
  Arms: Prospective Experimental Group
Other: Early Mobilization — Patient transferred up to the chair (within 5-30 minutes of admission to the recovery room) based on nursing parameters and patient safety.
  Arms: Prospective Experimental Group
Other: Early PO Intake — Patient will be offered PO intake within 15-30 minutes of admission to the recovery room post-procedure based on nursing parameters and patient safety.
  Arms: Prospective Experimental Group

SUMMARY:
The purpose of this study is to compare an Enhanced Recovery Pathway to the current pre-operative/recovery practices of the endoscopy department on patient post-procedure outcomes.

DETAILED DESCRIPTION:
Every 4th to 5th patient that checks in to the endoscopy department for their procedure will be screened for eligibility requirements. If eligible for the study, the patient will be informed about the study and potential risks. All patients giving written informed consent will be enrolled into the enhanced recovery protocol (ERP) [nursing managed ERP: goal-directed fluid management (Lactated Ringer's Solution at 5mL/kg/hr), PONV prophylaxis for an apfel score of 2 or greater (ondansetron 4 mg IV), early mobilization up to chair (within 5-30 minutes of admission to the recovery room), and early PO intake within 15-30 minutes of admission to the recovery room post-procedure] for their procedure.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient colonoscopy under moderate sedation
* Colonoscopy Indications: Screening

Exclusion Criteria:

* More than one sedation procedure scheduled same day
* Allergy to ondansetron
* Past PONV requiring scopolamine patches
* Diagnoses: ESRD, heart failure, cirrhosis, long QT syndrome
* Patients requiring fluid restrictions, such as dialysis patients
* Post-procedure NPO requirements, such as procedure-related NPO status (stent placement, pneumatic dilation, etc.) or second procedure in another location
* High Fall Risk Patients
* Adults unable to consent
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
To compare recovery time stamps before and after implementing a modified ERAs for endoscopy patients in the recovery period. | 1-2 hours
  We will compare mean recovery times between control and intervention groups using analysis of variance (ANOVA).
To compare the incidence of postoperative nausea and vomiting before and after implementing a modified ERAs for endoscopy patients in the recovery period. | 1-2 hours
  We will perform a Chi-square analysis for presence or absence of nausea and/or vomiting in the recovery period (measured by: administration of anti-emetic, documentation on N/V flowchart, and/or documentation in nursing narrative note) between control and intervention groups.

SECONDARY OUTCOMES:
To compare patient satisfaction scores before and after implementing a modified ERAs for endoscopy patients in the recovery period. | 15 minutes
  We will perform a t-test of patient satisfaction scores (Press Ganey scores) between control and intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Maeder, PhD, Principal Investigator — Northwestern Medicine
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alghanem SM, Massad IM, Rashed EM, Abu-Ali HM, Daradkeh SS. Optimization of anesthesia antiemetic measures versus combination therapy using dexamethasone or ondansetron for the prevention of postoperative nausea and vomiting. Surg Endosc. 2010 Feb;24(2):353-8. doi: 10.1007/s00464-009-0567-3. Epub 2009 Jun 11. PMID 19517165
- [Background] Amornyotin S. Sedation-related complications in gastrointestinal endoscopy. World J Gastrointest Endosc. 2013 Nov 16;5(11):527-33. doi: 10.4253/wjge.v5.i11.527. PMID 24255744
- [Background] Brown JK, Singh K, Dumitru R, Chan E, Kim MP. The Benefits of Enhanced Recovery After Surgery Programs and Their Application in Cardiothoracic Surgery. Methodist Debakey Cardiovasc J. 2018 Apr-Jun;14(2):77-88. doi: 10.14797/mdcj-14-2-77. PMID 29977464
- [Background] Apfel CC, Korttila K, Abdalla M, Kerger H, Turan A, Vedder I, Zernak C, Danner K, Jokela R, Pocock SJ, Trenkler S, Kredel M, Biedler A, Sessler DI, Roewer N; IMPACT Investigators. A factorial trial of six interventions for the prevention of postoperative nausea and vomiting. N Engl J Med. 2004 Jun 10;350(24):2441-51. doi: 10.1056/NEJMoa032196. PMID 15190136
- [Background] Ellett ML. Review of propofol and auxiliary medications used for sedation. Gastroenterol Nurs. 2010 Jul-Aug;33(4):284-95; quiz 296-7. doi: 10.1097/SGA.0b013e3181eac371. PMID 20679780
- [Background] Crenshaw JT, Winslow EH. Preoperative fasting: old habits die hard. Am J Nurs. 2002 May;102(5):36-44; quiz 45. doi: 10.1097/00000446-200205000-00033. PMID 12006853
- [Background] Gan TJ. Postoperative nausea and vomiting--can it be eliminated? JAMA. 2002 Mar 13;287(10):1233-6. doi: 10.1001/jama.287.10.1233. No abstract available. PMID 11886298
- [Background] Joliat GR, Ljungqvist O, Wasylak T, Peters O, Demartines N. Beyond surgery: clinical and economic impact of Enhanced Recovery After Surgery programs. BMC Health Serv Res. 2018 Dec 29;18(1):1008. doi: 10.1186/s12913-018-3824-0. PMID 30594252
- [Background] Lichtenstein GR, Cohen LB, Uribarri J. Review article: Bowel preparation for colonoscopy--the importance of adequate hydration. Aliment Pharmacol Ther. 2007 Sep 1;26(5):633-41. doi: 10.1111/j.1365-2036.2007.03406.x. PMID 17697197
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Saraghi M. Intraoperative Fluids and Fluid Management for Ambulatory Dental Sedation and General Anesthesia. Anesth Prog. 2015 Winter;62(4):168-76; quiz 177. doi: 10.2344/0003-3006-62.4.168. PMID 26650497
- [Background] Shaikh SI, Nagarekha D, Hegade G, Marutheesh M. Postoperative nausea and vomiting: A simple yet complex problem. Anesth Essays Res. 2016 Sep-Dec;10(3):388-396. doi: 10.4103/0259-1162.179310. PMID 27746521
- [Background] Som A, Bhattacharjee S, Maitra S, Arora MK, Baidya DK. Combination of 5-HT3 Antagonist and Dexamethasone Is Superior to 5-HT3 Antagonist Alone for PONV Prophylaxis After Laparoscopic Surgeries: A Meta-analysis. Anesth Analg. 2016 Dec;123(6):1418-1426. doi: 10.1213/ANE.0000000000001617. PMID 27870735
- [Background] Weinberg L, Faulkner M, Tan CO, Liu DH, Tay S, Nikfarjam M, Peyton P, Story D. Fluid prescription practices of anesthesiologists managing patients undergoing elective colonoscopy: an observational study. BMC Res Notes. 2014 Jun 10;7:356. doi: 10.1186/1756-0500-7-356. PMID 24916073